CLINICAL TRIAL: NCT06913166
Title: A Modified Pilot Randomised Controlled Trial (RCT) on the Effectiveness of an Online Quiz Game to Promote Tobacco-Related Knowledge, Attitudes, and Behaviours Among Primary School Students
Brief Title: Effectiveness of an Online Quiz in Promoting Tobacco-Related Knowledge, Attitudes, and Behaviours Among Primary Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hong Kong Council on Smoking and Health (Other)
Responsible Party: Principal Investigator, Au Yeung, Shiu Lun Ryan, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: coshdrama2425
Record Dates: First submitted 2025-03-19; First posted 2025-04-06 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Tobacco Prevention
Keywords: tobacco cessation; literacy; non-pharmaceutical intervention; adolescents
MeSH Terms: conditions — Tobacco Use Cessation; Literacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Quiz related to tobacco topics (Experimental): Students will engage in an online quiz competition for 5 days on tobacco-related topics. Each day, students could answer a maximum of 10 questions.
  Interventions: Other: Online quiz competition
- Quiz related to healthy eating topics (Active Comparator): Students will engage in an online quiz competition for 5 days on healthy eating-related topics. Each day, students could answer a maximum of 10 questions.
  Interventions: Other: Online quiz competition

INTERVENTIONS:
Other: Online quiz competition — Students in the intervention and control arm will participate in an online quiz game on tobacco or diet related topics respectively. Each day, students could answer a maximum of 10 questions randomly selected from the respective pool of questions by the platform. The students logged onto the online platform and played the quiz competition on weekdays for 5 days.

SUMMARY:
The goal of this modified pilot RCT is to evaluate the effects of the intervention (online platform) on tobacco-related knowledge, attitudes and intentions on smoking among local primary 5-6 school students. The main questions it aims to answer are:

* Is the intervention effective in improving tobacco-related knowledge (including alternative smoking products (ASPs) and tobacco control development in the world and Hong Kong)?
* Is the intervention effective in improving tobacco-related attitudes and intentions (including ASPs and tobacco control development in the world and Hong Kong)?

Researchers will compare the questionnaire results from students to see if intervention groups (students doing tobacco-related questions on the online quiz platform) will have better tobacco-related knowledge, higher anti-tobacco attitudes and lower intention to smoke.

ELIGIBILITY:
Inclusion Criteria:

* Primary 5-6 students from local primary schools
* Able to read and communicate in Chinese
* Have a digital device for online access to the quiz game at home

Exclusion Criteria:

* None

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 700 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of intervention on tobacco-related knowledge (including ASPs and tobacco control development in the world and Hong Kong) | Right before the intervention and at 8-12th days
  Students reported their opinions towards 5 statements in pre and post tests: [Pre-test] 1) Smoking causes wrinkles to form on the skin; 2) Third-hand smoke can remain on surfaces for weeks; 3) E-cigarettes can help with smoking cessation; 4) Tobacco companies aim to prevent teenagers from smoking; 5) The Hong Kong government has already banned the sale of e-cigarettes.
  [Post-test]
  1) Smoking can cause hair loss; 2) Opening windows or turning on a fan can eliminate the effects of thirdhand smoke; 3) E-cigarettes avoid the problem of secondhand smoke; 4) Tobacco companies hire influencers to promote tobacco products; 5) The Hong Kong government has already banned the sale of heated tobacco products.
  Students' knowledge will be assessed using a 5-point Likert scale, with each item rated on a 5-point Likert scale ranging from 1 (Strongly disagree) to 5 (Strongly agree). Item scores will be recoded as appropriate, so that higher scores consistently reflect better knowledge.
Effectiveness of intervention on tobacco-related attitudes (including ASPs and tobacco control development in the world and Hong Kong) | Right before the intervention and at 8-12th days.
  Students will report their opinions towards 5 statements: 1) Smoking is a selfish behavior; 2) I hope to avoid exposure to secondhand smoke; 3) Vaping is a trend.; 4) Tobacco companies use different methods to attract people to smoke; 5) The government should prohibit people from smoking while walking.
  Students' attitudes will be assessed using a 5-point Likert scale, with each item rated on a 5-point Likert scale ranging from 1 (Strongly disagree) to 5 (Strongly agree). Item scores will be recoded as appropriate, so that higher scores consistently reflect more negative attitudes.
Effectiveness of intervention on tobacco-related intentions (including ASPs and tobacco control development in the world and Hong Kong) | Right before the intervention and at 8-12th days.
  Students were asked: If one of your good friends offers you a traditional cigarette, e-cigarette or heated tobacco product, ask you to have a few puffs, and no one will know about this as no more smoking in the future. Will you use them?
  Students' intention will be assessed using a 5-point Likert scale, with each item rated on a 5-point Likert scale ranging from 1 (Definitely no) to 5 (Definitely yes). Lower scores indicate a lower intention to use ASPs.

SECONDARY OUTCOMES:
Effectiveness of intervention on SHS and THS exposure at home | Right before the intervention and at 8-12th days.
  Students were asked: In the past 7 days, how many days (0-7) 1) was someone smoking next to you when you were at home? 2) do you smell secondhand smoke drifting in from outside when you were at home? 3) was someone smoking next to you when you were outside home? 4) you can smell cigarette smoke on objects or people when you are at home and no one is smoking, and you don't see any smoke?
  Each item was rated on an 8-point scale ranging from 0 (0 days) to 7 (7 days), with higher scores indicating more frequent exposure to secondhand smoke (i.e., a worse outcome).
Effectiveness of intervention on tobacco use | Right before the intervention and at 8-12th days.
  Students were asked: 1) Which of the following tobacco products have you ever used? 2) In the past 30 days, which of the following tobacco products have you used?
Adherence to the 5-day intervention | At 8-12th days
  Students will report their adherence to the 5-day intervention. This information will be extracted directly from online quiz log of the participants via the backend of the system.
Satisfaction of students and parents towards intervention | From 2-8 weeks after the completion of the post-questionnaire
  These will be assessed using a qualitative interview for a subset of the participants and their family (10 students and parents)

CONTACTS AND LOCATIONS:
Overall Officials: Shiu Lun Ryan Au Yeung, Principal Investigator — School of Public Health, The University of Hong Kong
Locations (1):
- Local primary schools, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the results in this article, including text, tables, figures, and appendices, along with the study protocol and statistical analysis plan, will be available for sharing. Data access will be granted starting three months after publication and will remain available for up to five years. Researchers with a methodologically sound proposal aligned with the approved study objectives may request access by contacting the principal investigator(PI) (Ryan Au Yeung) at ayslryan@hku.hk. Approved data requestors will be required to sign a data-access agreement.
Supporting Information: Study Protocol
Time Frame: Starting three months after publication and will remain available for up to five years.
Access Criteria: Researchers with a methodologically sound proposal aligned with the approved study objectives may request access by contacting the PI (Ryan Au Yeung) at ayslryan@hku.hk. Approved data requestors will be required to sign a data-access agreement.